CLINICAL TRIAL: NCT04626115
Title: Diagnostic Performance of Sonazoid Contrast-enhanced Ultrasound in Renal Tumors
Brief Title: Diagnostic Value of Sonazoid Contrast-enhanced Ultrasound in Renal Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Diagnostic performance of Sonazoid contrast-enhanced ultrasound in renal tumors, Chinese PLA General Hospital
Other Study IDs: S2020-300-2
Record Dates: First submitted 2020-09-29; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Contrast Enhanced Ultrasound
Keywords: kidney

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence and mortality of renal cell carcinoma are increasing year by year. Contrast-enhanced ultrasound is helpful for early diagnosis and treatment to renal tumor, and is of great importance to distinguish benign from malignant and clinical stages

DETAILED DESCRIPTION:
The morbidity of renal cell carcinoma is only lower to prostate cancer and bladder cancer in urinary tumor, and the mortality rate is up to 40%. At present, diagnostic techniques such as ultrasonography, CT examination and MRI examination are widely used in Clinical practice, which greatly improves the detection rate of asymptomatic renal cell carcinoma. Compared with enhanced MRI and enhanced CT, contrast-enhanced ultrasound (CEUS) has outstanding advantages, including spatial, temporal and contrast resolution, continuous real-time visualization,. Sonazoid, the second generation ultrasound contrast agent, is composed of microbubbles containing chemically stable and insoluble perfluorobutane (PFB) gas and phosphatidylserine sodium hard shell (diameter 2-3μm) wrapped by outer layer. These microbubbles can generate stable nonlinear oscillation in low-power sound field, and generate echo at the second harmonic frequency of transmitted pulse. Sonazoid has the advantages of long-time development and good stability, which may improve the accuracy of distinguishing benign and malignant renal space-occupying lesions, especially small lesions. In addition, the characteristics of long-time development are also helpful to extract more imaging information to assist the clinical staging of renal tumors.

ELIGIBILITY:
Inclusion Criteria:

* (1) The subjects are able and willing to abide by the research procedure and sign the informed consent form; (2) The subjects who received CECT or CEMRI examination of renal tumor before the treatment; (4) Patients with no serious cardiovascular and cerebrovascular diseases; (5) Patients who intend to undergo biopsy or lesion resection；(6) aged 18 -85;。

Exclusion Criteria:

* (1) pregnant or lactating patients; (2) The subject has a history of allergy to eggs or egg products (i.e., general rash, dyspnea, swelling of mouth or throat, hypotension or shock, etc.); (3) It is known that the subject is allergic to perfluorobutane gas or any component of Sonazoid; (4) Patients who can't receive contrast MRI or enhanced CT examination.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The requirements of the case report form, the age, sex, smoking history, hypertension, diabetes, coronary heart disease, stroke history, general condition of the patients and physical examination results of the patients should be registered for outpatient or inpatient patients after obtaining the informed consent of the patients.
  If the patient is undergoing surgical treatment, record the operation mode, results and complications of the patient. Patients who need comprehensive treatment after operation should record the treatment measures and the name, usage and dosage of drugs.
  Contact information (fixed telephone or mobile phone) of at least two patients and their families should be obtained for future follow-up.
Sampling Method: Probability Sample
Enrollment: 223 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of contrast-enhanced ultrasound in renal tumor by Sonazoid. | 1 year
  Pathology as a gold standard, to compare the diagnostic performance between contrast-enhanced ultrasound and other contrast-enhanced imaging in renal tumor by Sonazoid.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No